CLINICAL TRIAL: NCT02260830
Title: Interventional, Open-label, Part Fixed Sequence, Part-randomised Study Investigating the Pharmacokinetic Properties of up to 6 Prototype Modified Release Tablet Formulations of Lu AF11167 in Healthy Young Subjects
Brief Title: Pharmacokinetic Properties of Various Modified Release Tablet Formulations of Lu AF11167
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15911A; 2013-004887-77 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-09 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Period A (Experimental): 1 reference treatment (2 mg Lu AF11167 immediate release hard capsule) + 5 different test prototype formulations of Lu AF11167
  Interventions: Drug: Lu AF11167
- Treatment Period B (Experimental): Food interaction and multiple dosing of Lu AF11167
  Interventions: Drug: Lu AF11167

INTERVENTIONS:
Drug: Lu AF11167

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic (PK) properties of various modified release tablet formulations of Lu AF11167 (Part A) and to investigate the pharmacokinetic (PK) properties of a modified release tablet formulation of Lu AF11167 in a fed and fasted state and following multiple dosing (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥18 and ≤45 years of age with a body mass index (BMI) of >18.5 and <30.0 kg/m2.
* Women of child-bearing potential will have a confirmed non-pregnant and non-lactating status.
* Other pre-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
PK parameters for Lu AF11167 estimated from the single dose treatment periods in Part A and B: Cmax, Frel, AUC0-inf, AUC0t, AUC%extr, CL/F, t½, tlag, tmax and Vz/F. | 0-48 hours
  Composite analysis
PK parameters for Lu AF11167 estimated from the multiple dose treatment period in Part B: AUC0-tau, AI (accumulation index), Cmax, Cpre, CL/F, t½, tmax and Vz/F. | Up to 60 hours post dose on day 7
  Composite analysis

SECONDARY OUTCOMES:
PK parameters for Lu AF36201 estimated from the single dose treatment periods in Part A and B: Cmax, AUC0-inf, AUC0-t, AUC%extr, t½, tlag and tmax, MR (metabolic ratio). | 0-48 HOurs
  Composite analysis
PK parameters for Lu AF36201 estimated from the multiple dose treatment period in Part B: AUC0-tau, AI, Cmax, Cpre, MR, t½ and tmax. | Up to 60 hours post dose day 7
  Composite analysis

OTHER OUTCOMES:
Number of adverse events | Up to 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via LundbeckClinicalTrials@Lundbeck.com, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom